CLINICAL TRIAL: NCT04652245
Title: Clinical Trial to Assess Onset of Action of Azelastine Hydrochloride and Fluticasone Propionate Nasal Spray Delivered in a Single Spray (Dymista) in the Treatment of Allergen-Induced Allergic Rhinitis Symptoms in Comparison to Placebo in an Environmental Exposure Unit (EEU)
Brief Title: Dymista Allergen Chamber - Onset of Action Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AZFL-AES-4-001; C1D00571 (Other: Cliantha Research, Canada)
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: The study will be a single-center, randomized, placebo-controlled, double-blind, and two-period cross-over trial.
Who Masked: Participant, Investigator
Masking Description: Blinding by overlabelling of Dymista and Placebo bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Dymista) and Treatment B (Placebo), separated by at least 14 days of wash-out period (Experimental): Fixed drug combination of Azelastine hydrochloride 137 μg / Fluticasone propionate 50 μg nasal spray and Placebo nasal spray
  Interventions: Drug: Treatment A (Dymista): Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 3; Drug: Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 5
- Treatment B (Placebo) and Treatment A (Dymista), separated by at least 14 days of wash-out period (Experimental): Placebo nasal spray and Fixed drug combination of Azelastine hydrochloride 137 μg / Fluticasone propionate 50 μg nasal spray
  Interventions: Drug: Treatment A (Dymista): Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 5; Drug: Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 3

INTERVENTIONS:
Drug: Treatment A (Dymista): Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 3 — Single dose, one spray in each nostril of Dymista nasal spray, approximately 137 μg of azelastine hydrochloride and 50 μg of fluticasone propionate per actuation, at Visit 3
  Arms: Treatment A (Dymista) and Treatment B (Placebo), separated by at least 14 days of wash-out period
Drug: Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 5 — Single dose, one spray in each nostril of Placebo nasal spray at Visit 5
  Arms: Treatment A (Dymista) and Treatment B (Placebo), separated by at least 14 days of wash-out period
Drug: Treatment A (Dymista): Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 5 — Single dose, one spray in each nostril of Dymista nasal spray, approximately 137 μg of azelastine hydrochloride and 50 μg of fluticasone propionate per actuation, at Visit 5
  Arms: Treatment B (Placebo) and Treatment A (Dymista), separated by at least 14 days of wash-out period
Drug: Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 3 — Single dose, one spray in each nostril of Placebo nasal spray, at Visit 3
  Arms: Treatment B (Placebo) and Treatment A (Dymista), separated by at least 14 days of wash-out period

SUMMARY:
This study is to assess the onset of action of fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray (Dymista) in treating the nasal symptoms of seasonal allergic rhinitis (SAR) induced by an allergen challenge in an Environmental Exposure Unit (EEU).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male or female subjects (childbearing and non-childbearing potential, non-childbearing potential defined as females with no menstruation for at least 1 year at screening and documented Follicle-Stimulating Hormone (FSH) > 35 IU/L) aged 18 to 55 years (inclusive) at screening.
3. History of SAR to ragweed pollen for at least the previous 2 ragweed pollen seasons.
4. Positive skin prick test (SPT) response to ragweed pollen (allergen induced wheal diameter at least 3 mm larger than the negative control). A test performed at Cliantha Research in the previous 12 months may be used to qualify the subject.
5. Willingness to complete all study visits.

   To be eligible for Visit 2 EEU, a subject must additionally comply with the following criteria:
6. Asymptomatic or with mild symptoms during the baseline recording of symptoms prior to start of the screening EEU (Visit 2):

   • Total Nasal Symptom Score (TNSS) ≤ 3/12 with the score for each symptom being less than 2.

   To be eligible for Visit 3, a subject must additionally comply with the following criteria during Visit 2 EEU:
7. Demonstrate adequate symptomology:

   • TNSS ≥ 6/12 on at least two Electronic Patient Data Acquisition Tablet (ePDAT TM) time point assessments during hours 0-2 in the EEU (Visit 2), with at least one occurring during the last two time points. Additionally, subjects will be required to meet a score of at least 2/3 for runny nose at least twice during hours 0-2 in the EEU, with at least one occurring during the last two time points.

   To be eligible for randomization (Visit 3), a subject must additionally comply with the following criteria:
8. Demonstrate adequate symptomology:

   * TNSS ≥ 6/12 on at least two ePDATTM time point assessments during hours 0-2 in the EEU (Visit 3), with at least one occurring during the last two time points. Additionally, subjects will be required to meet a score of at least 2/3 for runny nose at least twice during hours 0-2 in the EEU, with at least one occurring during the last two time points.
   * No evidence of complete nasal blockage on either one or both sides on anterior rhinoscopy within 30 minutes prior to dosing.

Exclusion Criteria:

Safety concerns:

1. History of allergic reaction to azelastine hydrochloride or fluticasone propionate or one of the excipients of the study treatments (e.g. benzalkonium chloride, phenylethyl alcohol, microcrystalline cellulose) or a component of the container.
2. History of anaphylaxis, cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, psychiatric, neurological, or other disease at screening that may affect subject safety during the study or evaluation of the study endpoints at the discretion of the Investigator and/or designee.
3. Subjects with a current diagnosis of asthma or subjects with measured Forced Expiratory Volume in 1 Second (FEV1) <75% of the predicted value using Global Lung Function Initiative set from 2012 for references.
4. Pregnant, breast-feeding or planning a pregnancy during the study and women of childbearing potential not using adequate contraception. Women of childbearing potential not abstinent or using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal Intrauterine Devices (IUDs), barrier methods, or tubal ligation started at least 4 weeks prior to screening.

   Lack of suitability for the study:
5. Previous and concomitant treatments: use of prohibited therapies (Antihistaminic agents, all presentations; Theophylline, all presentations; Cromolyn sodium, all forms; Nedocromil sodium; Salbutamol, all presentations; Leukotriene modifiers, all presentations; Corticosteroids (inhaled, oral, intravenous); Topical corticosteroids (ocular, intranasal); Corticosteroids (intramuscular or intra-articular); Decongestants, all forms; Immunotherapy; Systemic antibiotics; Tricyclic antidepressants and Monoamine Oxidase (MAO) inhibitors; Any cytochrome P450 3A4 inhibiting or inducing drug (e.g. ritonavir, cobicistat, ketoconazole, itraconazole, erythromycin, cimetidine, rifampicin, St. John's wort (Hypericum perforatum) etc.) not allowed within specific time frames prior to Screening and/or not allowed/allowed only with restrictions during the study, as specified in the study protocol; use of any medication considered to have an influence on the outcome of the study during the EEU session, at the discretion of the Investigator and/or designee.
6. Subjects with (expected) clinically relevant symptoms at the timing of the scheduled EEU assessments due to concomitant allergies, i.e. history of allergic response to the causative allergen, at the discretion of the Investigator. Subjects with a positive SPT for cats and/or dogs are acceptable if the subject avoids cats and/or dogs for the duration of the study.
7. Concomitant diseases: abnormalities during the screening visit (Visit 1) or Visit 2 that might interfere with study results as determined by the Investigator and/or designee.
8. Presence of a severely deviated septum, septal perforation, structural nasal defect or large nasal polyps causing obstruction as determined by the Investigator.
9. Acute conditions: any acute illness within 7 days prior to the screening visit (Visit 1) or Visit 2, including acute conjunctivitis or any other ocular infection, at the discretion of the Investigator and/or designee.
10. History of increased ocular pressure, glaucoma, cataracts, and/or central serous chorioretinopathy (CSCR).
11. Presence of or ongoing tuberculosis, untreated local or systemic fungal or bacterial infections, systemic viral or parasitic infections or ocular herpes simplex.
12. Recent nasal ulcers, mucosal erosion, nasal surgery, or nasal trauma, that might interfere with study results as determined by the Investigator and/or designee.
13. Exposure to chickenpox or measles within 4 weeks prior to the screening visit or during the study.
14. Acute or chronic sinusitis or non-allergic rhinitis, at the discretion of the Investigator and/or designee.
15. Exposure to another investigational product within the last 30 days prior to screening.
16. History of malignancy within the past five years, except for basal cell skin carcinomas that have been treated with no recurrence for at least 3 months.
17. Neurological or psychiatric disease or drug or alcohol abuse which would interfere with the subject's proper completion of the protocol assignment. Subjects with a positive urine drug screen will be excluded.
18. Subjects undergoing surgical procedures with general anaesthesia within 90 days prior to screening or who plan to undergo surgery/hospitalization during the study.

    Administrative reasons:
19. Vulnerable subjects (such as persons who are institutionalized).
20. Positive alcohol or drug test during screening visit (Visit 1)
21. Public health emergency (e.g. COVID-19): subjects not complying to Public health guidelines (e.g. self isolation etc.), at the discretion of the Investigator's and/or designee, or subjects with a positive COVID-test at Visit 2.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, Dr., Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment Administration Period 1: Treatment A or B at medical clinic, duration: 1 day; Wash out Period at home, duration: at least 14 days; Treatment Administration Period 2: Treatment B or A at medical clinic, duration: 1 day;
Period: Treatment Administration Period 1
Arm/Group | Treatment A (Dymista) and Treatment B (Placebo), Separated by at Least 14 Days of Wash-out Period | Treatment B (Placebo) and Treatment A (Dymista), Separated by at Least 14 Days of Wash-out Period
Started | 108 | 108
Completed | 108 | 108
Not Completed | 0 | 0
Period: Wash-Out Period
Arm/Group | Treatment A (Dymista) and Treatment B (Placebo), Separated by at Least 14 Days of Wash-out Period | Treatment B (Placebo) and Treatment A (Dymista), Separated by at Least 14 Days of Wash-out Period
Started | 108 | 108
Completed | 108 | 104
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Treatment Administration Period 2
Arm/Group | Treatment A (Dymista) and Treatment B (Placebo), Separated by at Least 14 Days of Wash-out Period | Treatment B (Placebo) and Treatment A (Dymista), Separated by at Least 14 Days of Wash-out Period
Started | 108 | 104
Completed | 108 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: FAS population includes all randomized patients, including subjects who received incorrect treatment, did not complete the study or did not comply to the protocol, and who were randomized but did not take any study medication
Groups:
- Entire Study Population (Crossover Design: Randomization to Dymista/Placebo or Placebo/Dymista): Fixed drug combination of Azelastine hydrochloride 137 μg / Fluticasone propionate 50 μg nasal spray and Placebo nasal spray
  Treatment A (Dymista): Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 3 OR Visit 5: Single dose, one spray in each nostril of Dymista nasal spray, approximately 137 μg of azelastine hydrochloride and 50 μg of fluticasone propionate per actuation, at Visit 3 OR Visit 5.
  Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 5 OR Visit 3: Single dose, one spray in each nostril of Placebo nasal spray at Visit 5 OR Visit 3.
Arm/Group | Entire Study Population (Crossover Design: Randomization to Dymista/Placebo or Placebo/Dymista)
Number analyzed (Participants) | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 216
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 186
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: American Indian or Alaska Native | 1
  Race, Customized: Asian | 41
  Race, Customized: Native Hawaiian or Other Pacific Islander | 0
  Race, Customized: Black or African American | 51
  Race, Customized: White | 117
  Race, Customized: Other | 6
Region of Enrollment [Number; unit: participants]
  Canada | 216
Height [Mean (Standard Deviation); unit: cm] | 169.7 (8.85)
Weight [Mean (Standard Deviation); unit: kg] | 79.38 (18.473)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.50 (5.817)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-assessed Instantaneous Total Nasal Symptom Score (TNSS) From Baseline Compared to Placebo
Description: FDA guideline defines onset of action as the first time point after initiation of treatment when the product demonstrated a greater change from baseline compared to placebo which proved durable.
  In this study, the first significant difference to placebo of TNSS was observed at 5 minutes time point (= onset of action).
  The TNSS is comprised of 4 symptoms from the nose, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TNSS contributes to a score ranging from 0 - 12.
Time Frame: 0 to 4 hours post application
Population: FAS (Full Analysis Set) population includes all randomized patients, including subjects who received incorrect treatment, did not complete the study or did not comply to the protocol, and who were randomized but did not take any study medication. Overall number of Participants Analyzed means the number of participants for whom the respective TNSS value at 5 min post-dose was available.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Treatment A (Dymista), Cross-over Design, Time-point 5 Min Post-dose (Onset of Action): Fixed drug combination of Azelastine hydrochloride 137 μg / Fluticasone propionate 50 μg nasal spray:
  Total Nasal Symptom Score (TNSS) difference to baseline after 5 min. post-dose
  Treatment A (Dymista) Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 3 OR Visit 5: Single dose, one spray in each nostril of Dymista nasal spray, approximately 137 μg of azelastine hydrochloride and 50 μg of fluticasone propionate per actuation, at Visit 3 OR Visit 5
- Treatment B (Placebo), Cross-over Design, Time-point 5 Min Post-dose (Onset of Action): Placebo nasal spray: Total Nasal Symptom Score (TNSS) difference to baseline after 5 min. post-dose
  Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 5 OR Visit 3: Single dose, one spray in each nostril of Placebo nasal spray at Visit 5 OR Visit 3
Arm/Group | Treatment A (Dymista), Cross-over Design, Time-point 5 Min Post-dose (Onset of Action) | Treatment B (Placebo), Cross-over Design, Time-point 5 Min Post-dose (Onset of Action)
Number analyzed (Participants) | 211 | 216
score on a scale | -1.37 (0.130) | -1.04 (0.128)
Statistical Analysis 1: Comparison: Treatment A (Dymista), Cross-over Design, Time-point 5 Min Post-dose (Onset of Action) vs Treatment B (Placebo), Cross-over Design, Time-point 5 Min Post-dose (Onset of Action); Test type: Superiority; p = 0.028, ANCOVA

2. Secondary Outcome: Change in Patient-assessed Instantaneous Total Ocular Symptom Score (TOSS) From Baseline Compared to Placebo
Description: FDA guideline defines onset of action as the first time point after initiation of treatment when the product demonstrated a greater change from baseline compared to placebo which proved durable.
  In this study, the first significant difference to placebo of TOSS was observed at 10 minutes time point (= onset of action).
  The TOSS is comprised of 3 symptoms from the eyes, each scored on a scale of 0 to 3 (0 = none and 3 = severe). The sum of the TOSS contributes to a score ranging from 0 - 9.
Time Frame: 0 to 4 hours post application
Population: FAS population includes all randomized patients, including subjects who received incorrect treatment, did not complete the study or did not comply to the protocol, and who were randomized but did not take any study medication. Overall number of Participants Analyzed means the number of participants for whom the respective TOSS value at 10 min post-dose was available.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Treatment A (Dymista), Cross-over Design, Time-point 10 Min Post-dose (Onset of Action): Fixed drug combination of Azelastine hydrochloride 137 μg / Fluticasone propionate 50 μg nasal spray:
  Total Ocular Symptom Score (TOSS) difference to baseline after 10 min. post-dose
  Treatment A (Dymista) Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 3 OR Visit 5: Single dose, one spray in each nostril of Dymista nasal spray, approximately 137 μg of azelastine hydrochloride and 50 μg of fluticasone propionate per actuation, at Visit 3 OR Visit 5
- Treatment B (Placebo), Cross-over Design, Time-point 10 Min Post-dose (Onset of Action): Placebo nasal spray: Total Ocular Symptom Score (TOSS) difference to baseline after 10 min. post-dose
  Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 5 OR Visit 3: Single dose, one spray in each nostril of Placebo nasal spray at Visit 5 OR Visit 3
Arm/Group | Treatment A (Dymista), Cross-over Design, Time-point 10 Min Post-dose (Onset of Action) | Treatment B (Placebo), Cross-over Design, Time-point 10 Min Post-dose (Onset of Action)
Number analyzed (Participants) | 211 | 215
score on a scale | -1.21 (0.104) | -0.87 (0.103)
Statistical Analysis 1: Comparison: Treatment A (Dymista), Cross-over Design, Time-point 10 Min Post-dose (Onset of Action) vs Treatment B (Placebo), Cross-over Design, Time-point 10 Min Post-dose (Onset of Action); Test type: Superiority; p = 0.008, ANCOVA

ADVERSE EVENTS:
Time Frame: In this study, the adverse event (AE) collection period began at the signing of informed consent and continued until 5 to 7 days after the last dose of study medication. AEs occurring during this period needed to be reported.
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product including an abnormal laboratory or physical findings, symptoms, or disease (new or exacerbated)) temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Subjects have been routinely queried in regard to the presence or absence of adverse events using open ended questions. Any AEs have been documented in the subject's eCRF.
Groups:
- Treatment A (Dymista), Cross-over Design: Fixed drug combination of Azelastine hydrochloride 137 μg / Fluticasone propionate 50 μg nasal spray:
  Treatment A (Dymista) Fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray at Visit 3 OR Visit 5: Single dose, one spray in each nostril of Dymista nasal spray, approximately 137 μg of azelastine hydrochloride and 50 μg of fluticasone propionate per actuation, at Visit 3 OR Visit 5
- Treatment B (Placebo), Cross-over Design: Placebo nasal spray
  Treatment B (Placebo): Nasal spray with no active dose (Dymista vehicle) at Visit 5 OR Visit 3: Single dose, one spray in each nostril of Placebo nasal spray at Visit 5 OR Visit 3
- Not Dedicated to Any Treatment Group: AEs not considered Treatment Emergent Adverse Events (not occurring in the period from administration of study medication until 5 days (120 h) thereafter)
Arm/Group | Treatment A (Dymista), Cross-over Design | Treatment B (Placebo), Cross-over Design | Not Dedicated to Any Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/216 | 0/216
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/216 | 0/216
Other Adverse Events (participants affected / at risk) | 2/212 | 6/216 | 9/216
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (Dymista), Cross-over Design (N=212) | Treatment B (Placebo), Cross-over Design (N=216) | Not Dedicated to Any Treatment Group (N=216)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 6 (6)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is an employee of the CRO (Contract Research Organization) and disclosure restrictions are specified by the agreement with the CRO. CRO shall not publish any study results without the prior written express consent of the Sponsoring company. In the event that such consent is given the Sponsoring company shall have 90 days from receipt of the proposed publication to review and comment. The Sponsor can require changes to the publication and delay of 90 days to the publication.

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04652245/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04652245/SAP_001.pdf